CLINICAL TRIAL: NCT03738176
Title: The Efficacy of Topical Sesame Oil in Orabase Versus Topical Triamcinolone in Orabase on Oral Lichen Planus and Salivary Level of Oxidative Stress Biomarker, Malondialdehyde [MDA] : Randomized Clinical Trial (RCT)
Brief Title: The Efficacy of Topical Sesame Oil Versus Topical Triamcinolone on Oral Lichen Planus and Salivary Level of Oxidative Stress Biomarker [MDA]
Acronym: (MDA)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mona Taha Mohammed MD (Other)
Responsible Party: Sponsor-Investigator, Mona Taha Mohammed MD, clinical researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2:5:1
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2018-11

CONDITIONS: Oral Lichen Planus
Keywords: Oral lichen planus; sesame oil; corticosteroid; MDA
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Sesame Oil; Triamcinolone; Orabase

STUDY DESIGN:
Intervention Model Description: sesame oil in orabase(80 gm CMC -20 gm sesame oil)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sesame oil in orabase (Experimental): 20 gm sesame oil-80 gm CMC 3 times per day for one month
  Interventions: Drug: Sesame Oil
- triamcinolone in orabase (Active Comparator): 140 gm triamcinolone-50 gm Na CMC 3 times per day for one month
  Interventions: Drug: triamcinolone in orabase

INTERVENTIONS:
Drug: Sesame Oil — Sesame oil(80 gm NaCMC-20 gmSesame oil)
  Other Names: sesame oil gel
  Arms: sesame oil in orabase
Drug: triamcinolone in orabase — triamcinolone 140 gm-Na CMC 50 gm
  Other Names: kenacorte
  Arms: triamcinolone in orabase

SUMMARY:
use seseme oil and corticosteroid topically for two groups

DETAILED DESCRIPTION:
* The enrolled patients will be divided randomly into two groups.
* Test group will receive topical sesame oil (3 times /day after eating) for a month.
* Control group will receive topical corticosteroid (3 times /day after eating) for a month.
* Assessment of the appearance score and severity of pain as well as the clinical parameter outcome will be done at baseline and at the end of two and four weeks and will be recorded in the patients' questionnaires & by clinical sign score . MDA will be measured at the baseline & at the end of four weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be clinically diagnosed as having atrophic &/or erosive oral lichen planus.

  * Patients with no history of taking topical corticosteroids for the last 2 months and systemic corticosteroid for the last 6 months
  * Patients who agree to take medication and follow up .

Exclusion Criteria:

* Pregnant and lactating ladies.

  * Patients with history of topical steroids during last 2 months & systemic steroids during last 6 months.
  * Patients with recent dental filling associated with the lesion or associated with recent drug administration.
  * Patient with history of diabetes or hypertension or those with positive HCV ab or HBs Ag.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-16 (Estimated); Primary Completion 2020-11-16 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
pain intensit measure | 4 weeks
  measured by visual analogue scale where0 no pain and 10 sever pain
reduction of clinical signs measure | 4 weeks
  Thongprasom Score 5 = white striae with erosive area = 1 cm2 Score 4 = white striae with erosive area < 1 cm2 Score 3 = white striae with erosive area > 1 cm2 Score 2 = white striae with atrophic area < 1 cm2 Score 1 = mild white striae only Score 0 = no lesion normal

SECONDARY OUTCOMES:
Salivary level of oxidative stress biomarker (MDA) | 4 weeks
  measured by reaction with thiobarbituric acid (TBA)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Taha Mohammed Ahammed, MD, Principal Investigator — Cairo U

IPD SHARING:
Plan to Share IPD: No